CLINICAL TRIAL: NCT00881582
Title: Peginterferon Alfa-2a Plus Ribavirin Combination Treatment in Chronic Hepatitis C Post-Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz Medical City (Other Government)
Collaborators: Riyadh Military Hospital (Other); King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Faisal M Sanai, Consultant Hepatologist & Liver Transplant Physician, King Abdulaziz Medical City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMH-01-09
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Hepatitis C; Renal Transplant
Keywords: Hepatitis c; Renal transplantation; Pegylated interferon
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pegylated interferon alfa-2a plus ribavarin (Experimental): Pegylated interferon alfa-2a plus ribavarin for 48 weeks
  Interventions: Drug: Pegylated interferon alfa-2a plus ribavarin

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a plus ribavarin — PEG-interferon alfa-2a and ribavirin. Pegylated interferon alfa-2a - standard dose; plus ribavirin - standard dose (determined by creatinine clearance); for 24 to 48 weeks (genotypes 1 & 4: 48 weeks; genotypes 2 & 3: 24 weeks)
  Other Names: Pegasys®, F. Hoffman-LaRoche; Copegus®, F. Hoffman-LaRoche

SUMMARY:
There is a distinct lack of published literature on the effect of combination treatment of PEG-interferon and ribavirin on post-renal transplantation hepatitis C virus (HCV) patients. Small case series have been published utilizing conventional interferon and/or ribavirin and the available data is extremely preliminary in nature. A small retrospective series of patients treated with Pegylated interferon and ribavirin published recently suggests that the treatment may be safe and efficacious. Unpublished reports from a few centers within Saudi Arabia also suggest a good safety profile and reasonable efficacy from this form of combination treatment.

The investigators aim to prospectively study the safety and efficacy of PEG-interferon and ribavirin combination therapy in post-renal transplant HCV-infected patients. Towards this 40 patients with histological evidence of liver disease will be recruited and the efficacy of the above medications studied.

The proposed study aims to evaluate the efficacy and safety of PEG-interferon and ribavirin combination therapy in the treatment of chronic HCV in renal transplant patients in a way that will allow management of such patients in an optimized manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male and female, aged 18 - 68 years
* Post renal transplant patients exceeding one year
* Anti-HCV (Abbott HCV EIA 2.0, Abbott Diagnostic, Chicago, IL) positive > 6 months AND/OR
* Detectable serum quantitative HCV-RNA (Cobas Amplicor HCV Monitor v2.0, Roche Molecular Systems, Pleasanton, CA) with lower limit of detection at 50 IU/mL
* Compensated liver disease with the following minimum hematologic and biochemical criteria:
* Hemoglobin > 10 g/dL
* WBC > 3000/mm3 ; granulocyte count > 1,500/mm3
* Platelet count > 75,000/mm3
* Albumin within normal limits
* TFT within normal limits
* ANA < 1:320
* Ultrasound of the liver obtained within the preceding 6 months of study entry
* Liver biopsy prior to entry confirming a histological diagnosis consistent with HCV necroinflammatory score (METAVIR) > 1, and fibrosis score >/= 2.

Exclusion Criteria:

* Previous treatment with interferon and / or Ribavirin - based therapy for chronic hepatitis C
* Co-infection with HBV or HIV
* Chronic alcohol abuse (daily consumption > 20 g/day)
* Autoimmune or metabolic liver disease liver disease
* Active drug-induced hepatitis or HAV
* Decompensated liver disease (Child-Pugh classification B or C) including a past history of decompensation
* Variceal bleeding
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration) or clinically relevant ophthalmological disorder due to diabetes mellitis or hypertension
* Neoplastic disease
* Patients with a value of alpha-fetoprotein >100 ng/mL will be excluded from the study until imaging studies confirm the absence of HCC. Presence of HCC, as determined by other means will also exclude the patient from histological sampling.
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (40 g/L) (as may be seen with ribavirin therapy) would not be well-tolerated
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* Evidence of drug abuse (including excessive alcohol consumption) within one year of study entry
* Current pregnancy, ongoing breast feeding or unwilling to have contraception
* Bleeding or clotting diatheses
* Recent history of renal allograft rejection (< 6 months)
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.
* History of organ transplantation, other than kidney, with an existing functional graft.
* Patients requiring dialysis or in whom dialysis is impending.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response | At 24 weeks post completion of treatment

SECONDARY OUTCOMES:
Adverse event rate and number of cases of graft rejection | Assessment at 4, 12, 24 and 48 weeks on treatment, and 24 weeks post completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Faisal M Sanai, MBBS, MD, Principal Investigator — Riyadh Military Hospital
Locations (2):
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Centre, Riyadh
  - Riyadh Military Hospital, Riyadh

REFERENCES:
- [Derived] Sanai FM, Mousa D, Al-Mdani A, Al-Shoail G, Al-Ashgar H, Al Meshari K, Al-Qahtani A, Saadeh M, Bzeizi KI, Aleid H. Safety and efficacy of peginterferon-alpha2a plus ribavirin treatment in renal transplant recipients with chronic hepatitis C. J Hepatol. 2013 Jun;58(6):1096-103. doi: 10.1016/j.jhep.2013.02.004. Epub 2013 Feb 18. PMID 23428875